CLINICAL TRIAL: NCT01205646
Title: Pilot Trial to Evaluate Change in Positron Emission Tomography Scanning (PET) as a Surrogate for Zoledronate (Zometa) Efficacy in Patients With Metastatic Prostate Cancer
Brief Title: PET Scanning to Evaluate Zoledronate Efficacy in Metastatic Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ulka Vaishampayan, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: WSU 2006-066
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Results first posted 2014-06-06 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; metastatic; zoledronate; zometa
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Zoledronic Acid; Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Zometa & PET Scans (Experimental): Zoledronate therapy & PET scan ;2 scans [about 1-2 weeks apart] will be obtained over a period of 2 weeks pretherapy to confirm reproducibility, Bone scan (within 4 weeks prior to registration), bone turnover markers, and PSA will be obtained pretherapy. After that, Zometa will be administered at a dose of 4mg IV over 15 minutes. A third PET scan will be obtained within 1-2 weeks after Zometa administration.
  Interventions: Drug: zoledronate therapy; Device: PET Scan

INTERVENTIONS:
Drug: zoledronate therapy — Zometa will be administered at a dose of 4mg IV over 15 minutes. A third PET scan will be obtained within 1-2 weeks after Zometa administration. Intravenous (through a vein in the arm) infusion every four weeks. Dose will be determined by kidney function.
  Other Names: Zometa
Device: PET Scan — 2 scans [about 1-2 weeks apart] will be obtained over a period of 2 weeks pretherapy to confirm reproducibility.A third PET scan will be obtained within 1-2 weeks after Zometa administration.

SUMMARY:
The primary goal for this trial is to assess the change in PET scans with the administration of zoledronate (bisphosphonate) therapy in patients with metastatic prostate cancer. It has been established that zoledronate therapy may play a role in delaying and reducing the incidence of skeletal events. Researchers propose to evaluate the change in the uptake value of FMAU PET scan after the zoledronate therapy. It has been demonstrated that FMAU PET scans can successfully demonstrate and detect bony metastatic sites in prostate cancer.

In addition, investigators would like to evaluate the change in the level of the prostate-specific antigen (PSA) in the patient as well as outcome of bone scans.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of prostate cancer
* Evidence of metastatic disease by radiologic criteria
* Bone scan within 4 weeks of starting therapy
* Creatinine within 2 weeks of registration, calculated creatinine clearance > 60ml/min.
* Minimum life expectancy of 6 months
* Willingness to have pre-therapy PET scans performed within 2 weeks after registration and post therapy PET scan performed within 1 week after dose of Zometa (a total of 3 PET scans required)
* Calculated creatinine clearance > 50ml/min.
* No prior Zoledronate therapy
* Patients must have disease progression despite testosterone suppression (level<50ng/ml); progression can be by rising PSA ( at least 2 values at least 2 weeks apart) or by new lesions on scans or progression of existing lesions on CT scan.
* No concomitant systemic therapy for metastatic prostate cancer is allowed except LHRH analogue should be continued if necessary to maintain testosterone suppression.
* No concomitant radiation therapy
* Prior RT is allowed if completed at least 2 weeks prior to registration.
* Presence of measurable or evaluable disease
* If RT has been administered, disease outside the RT port is required.
* Willingness to sign informed consent.
* Registration and willingness to sign informed consent for separate PET protocol 2335 that describes the PET scan procedure.
* Patients must have good oral hygiene which includes having a recent dental evaluation

Exclusion Criteria:

* Patients who are unable to swallow
* Patients with dental cavities that are likely to need dental extraction or root canal treatment as management

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-09; Primary Completion 2013-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulka N. Vaishampayan, M.D., Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (2):
- United States (2):
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Karmanos Cancer Institute Weisberg Cancer Treatment Center, Farmington Hills, Michigan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zometa & PET Scans
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Zometa & PET Scans
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.09 (4.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: PET Response Rate in Metastatic Prostate Cancer Patients Treated With Zoledronate Therapy.
Description: PET response rate was pre-defined in Section 5.0 of the protocol based on the magnitude of change in the mean standardized uptake value (SUVmean), which is measured at each PET scan. Specifically, a decline in SUVmean of at least 15% pre/post Zometa was taken as evidence of a "PET response". Per the protocol, Scan 2 was used as the pre-Zometa measure of SUVmean, and Scan 3 (1-2 weeks later) was used as the post-Zometa measure of SUVmean.
Time Frame: Within 3 weeks
Measure: Number (90% Confidence Interval); unit: Proportion of participants with response
Arm/Group | Zometa & PET Scans
Number analyzed (Participants) | 11
Proportion of participants with response | .091 [.021 to .323]

2. Secondary Outcome: The Change in PSA After Zoledronate Therapy
Description: The change in PSA after zoledronate therapy using per cent change.
Time Frame: Four weeks after initiating Zoledronate therapy
Population: All patients who had their PSA measured both before and after therapy.
Measure: Median (Full Range); unit: percentage of change in PSA
Arm/Group | Zometa & PET Scans
Number analyzed (Participants) | 10
percentage of change in PSA | 38.99 [-34.09 to 408.89]

3. Secondary Outcome: Change in Bone Scans
Description: Change in bone scans using per cent change in SUVmax.
Time Frame: Four weeks after initiating zoledronate therapy
Population: Sample population
Measure: Median (Full Range); unit: percentage of change of SUVmax
Arm/Group | Zometa & PET Scans
Number analyzed (Participants) | 11
percentage of change of SUVmax | -10.08 [-43.84 to 54.78]

4. Secondary Outcome: Changes in Bone Turnover Markers
Description: Changes in bone turnover markers using per cent change of BSAP and NTx
Time Frame: Four weeks after initiating zoledronte therapy
Population: Patients who had both pre-treatment and post-treatment measures of BSAP and NTx.
Measure: Median (Full Range); unit: percentage of change in bio-marker
Arm/Group | Zometa & PET Scans
Number analyzed (Participants) | 11
percentage of change in bio-marker
  BSAP | -1.66 [-29.80 to 44.08]
  NTx | -68.18 [-82.35 to -50.00]

ADVERSE EVENTS:
Arm/Group | Zometa & PET Scans
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 3/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zometa & PET Scans (N=11)
Myalgias (Musculoskeletal and connective tissue disorders) | 2 (2)
Chills (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No